CLINICAL TRIAL: NCT01325714
Title: Preventing Aggression in Veterans With Dementia
Acronym: PAVeD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 09-351
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Dementia; Aggression; Pain
MeSH Terms: conditions — Dementia; Aggression; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: PAVeD Intervention (Experimental): In the experimental arm, the caregiver will receive six to eight 45-minute visits to teach caregiver about pain and memory problems. The person with dementia will also be able to learn from these visits. These visits will take place over three months.
  Interventions: Behavioral: PAVeD Intervention
- Arm 2: Enhanced Usual Care (Active Comparator): In the comparison arm, the caregiver will receive information in the mail about memory problems and pain; and the caregiver will receive eight short telephone calls to check on how the person with dementia is doing.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: PAVeD Intervention — In the PAVeD Intervention, the caregiver will receive six to eight 45-minute visits to teach caregiver about pain and memory problems. The person with dementia will also be able to learn from these visits. These visits will take place over three months.
  Arms: Arm 1: PAVeD Intervention
Behavioral: Enhanced Usual Care — In Enhanced Usual Care, the caregiver will receive information in the mail about memory problems and pain; and the caregiver will receive eight short telephone calls to check on how the person with dementia is doing.
  Primary Care providers will be notified through electronic medical records about any significant behavioral problems or pain.
  Arms: Arm 2: Enhanced Usual Care

SUMMARY:
This study tests whether education about memory and pain might help to prevent aggression in persons with dementia who have pain. The overall goal of this intervention is to reduce the risk of aggressive behavior by improving several areas of patient life that are known causes of aggression: pain, depression, lack of pleasurable activities, caregiver stress and difficulty in caregiver-patient communication.

DETAILED DESCRIPTION:
Dementia is known primarily for its effects on memory, however, eighty percent of persons with dementia also have behavioral disturbances. This is often not addressed, leading to increased use of nursing homes, higher incidence of injury (both patient and caregiver) and the use of tranquilizing medications. Pain is one of the strongest predictors of aggression. The prevalence of pain in persons with dementia is known to be about 50%. Untreated pain is associated with significant negative outcomes, including increased health care use, inactivity and isolation. The investigators aim to determine whether outcome differences exist between active intervention and control conditions in relation to the occurrence of aggressive behavior, pain and depression, and its impact on pleasant activities, caregiver burden, quality of caregiver-patient relationship, antipsychotic use, health-service use, injuries to patient and caregiver, and nursing home placement. The active intervention, Preventing Aggression in Veterans with Dementia (PAVeD), is a family caregiver-focused, home-based intervention that uses psychoeducational and behavioral approaches to help reduce the risk of aggressive behavior in persons with dementia. The objective of PAVeD is to improve several areas of patient life that are known causes of aggression: pain and distress (including mood problems), lack of pleasurable activities, and difficulty in patient-caregiver communication that may negatively affect relationship quality and caregivers' recognition of pain.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to participate in the study if they meet the following criteria:

* have a documented diagnosis of dementia
* receive primary care from the VA
* reside outside a long-term care facility
* live within 45 minutes of the MEDVAMC
* have mild-to-moderate dementia
* have no history of aggression in the past year
* have no evidence of aggression on the CMAI at baseline (i.e., do not score 2 or higher on both frequency and disruptiveness for any of 13 behaviors listed).
* have a caregiver who is directly involved with the patient:

  * at least 8 hours per week
  * sees the patient at least twice a week
  * and speaks English
* report clinically significant pain (either directly or through the caregiver as a proxy)

Exclusion Criteria:

Patients will be excluded if they have had history of aggression in the past year

* The investigators will administer the aggression subscale of the Cohen-Mansfield Agitation Inventory (CMAI)
* Aggression will be considered present if any of the following items are endorsed as having occurred over the prior year:

  * spitting
  * cursing/verbal aggression
  * hitting
  * kicking
  * grabbing
  * pushing
  * throwing
  * biting
  * scratching
  * hurting self/others
  * tearing things/destroying property
  * making inappropriate verbal sexual advances
  * or making inappropriate physical sexual advances

Participants that scored 2 or higher for both frequency and disruptiveness on any of the 13 behaviors listed on the CMAI at baseline were considered aggressive and were excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2011-05; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Kunik, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fowler JH, Dannecker K, Stanley M, Wilson N, Snow AL, Kunik ME. Preventing aggression and other secondary features of dementia in elderly persons: Three case studies. Bull Menninger Clin. 2015 Spring;79(2):95-115. doi: 10.1521/bumc.2015.79.2.95. PMID 26035086
- [Result] Bradford A, Shrestha S, Snow AL, Stanley MA, Wilson N, Hersch G, Kunik ME. Managing pain to prevent aggression in people with dementia: a nonpharmacologic intervention. Am J Alzheimers Dis Other Demen. 2012 Feb;27(1):41-7. doi: 10.1177/1533317512439795. PMID 22467413
- [Result] Breland JY, Barrera TL, Snow AL, Sansgiry S, Stanley MA, Wilson N, Amspoker AB, Kunik ME. Correlates of pain intensity in community-dwelling individuals with mild to moderate dementia. Am J Alzheimers Dis Other Demen. 2015 May;30(3):320-5. doi: 10.1177/1533317514545827. Epub 2014 Aug 7. PMID 25107934
- [Result] Li J, Snow AL, Wilson N, Stanley MA, Morgan RO, Sansgiry S, Kunik ME. The Quality of Pain Treatment in Community-Dwelling Persons with Dementia. Dement Geriatr Cogn Dis Extra. 2015 Dec 5;5(3):459-70. doi: 10.1159/000441717. eCollection 2015 Sep-Dec. PMID 26955380
- [Derived] Amspoker AB, Snow AL, Renn BN, Block P, Pickens S, Morgan RO, Kunik ME. Patient Versus Informal Caregiver Proxy Reports of Pain Interference in Persons With Dementia. J Appl Gerontol. 2021 Apr;40(4):414-422. doi: 10.1177/0733464820902632. Epub 2020 Feb 6. PMID 32026743

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: PAVeD Intervention: 106 caregivers were randomized to the PAVeD intervention. Five were excluded at baseline because of aggression. 101 caregivers were included in the primary analysis. Dyads assigned to PAVeD received 6 to 8 weekly sessions of 45-minute home visits. PAVeD consists of 4 weekly 45- minute "core" sessions ("Recognizing Pain"; "Recognizing and Responding to Pain and Distress"; "Enhancing Communication"; "Making Daily Activities More Pleasant and Enjoyable") and 2 of 4 elective sessions ("Medical Treatments and Talking to Your Doctor," "Rest and Relaxation Strategies," "Communication Problems and Challenges," and "Increasing Pleasant Activities"), chosen with the patient and/or caregiver through collaborative goal setting during the first session. The intervention includes didactics, skill-building, discussion, and role-playing guided by a clinician manual and caregiver workbook.
- Arm 2: Enhanced Usual Care: 107 caregivers were randomized to Enhanced Usual Care. Three were excluded at baseline because of aggression and two dropped out prior to baseline (one withdrew and one deceased). 102 caregivers were included in primary analysis. Dyads assigned to EU-PC received 8 weekly 15-minute phone calls to query symptom severity, ascertain needs for immediate psychiatric care, and provide minimal support. Primary care physicians of patients assigned to both groups received American Medical Association Continuing Medical Education print material on treating pain in older adults, as well as feedback progress notes documenting the PWD's level of pain and depression at baseline, 3 months, 6 months, and 12 months
Period: Overall Study
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Started | 101 | 102
3 Month Assessment | 82 | 86
6 Month Asessment | 75 | 82
12 Month Assessment | 67 | 71
Completed | 67 | 71
Not Completed | 34 | 31

BASELINE CHARACTERISTICS:
Population: We evaluated differences in demographics and baseline clinical characteristics between PAVeD and EU-PC subgroups using chi-square tests and independent samples t-tests. however, when distributional assumptions were violated, a non-parametric Fishers Exact or Wilcoxon Mann-Whitney U test was conducted.
Groups:
- Arm 2: Enhanced Usual Care: In the comparison arm, the caregiver will receive information in the mail about memory problems and pain; and the caregiver will receive eight short telephone calls to check on how the person with dementia is doing.
  Enhanced Usual Care: In Enhanced Usual Care, the caregiver will receive information in the mail about memory problems and pain; and the caregiver will receive eight short telephone calls to check on how the person with dementia is doing.
  Primary Care providers will be notified through electronic medical records about any significant behavioral problems or pain.
- Total: Total of all reporting groups
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care | Total
Number analyzed (Participants) | 101 | 102 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.21 (8.46) | 80.26 (8.00) | 79.24 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 101 | 98 | 199
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 47 | 47 | 94
  Black | 36 | 37 | 73
  Hispanic or Latino | 15 | 15 | 30
  Other | 3 | 3 | 6
Caregiver age (continuous) [Mean (Standard Deviation); unit: years] | 66.43 (12.54) | 65.69 (12.72) | 66.06 (12.61)
Caregiver gender (categorical) [Number; unit: participants]
  Males | 6 | 10 | 16
  Females | 95 | 92 | 187
Caregiver race/ethnicity (categorical) [Number; unit: participants]
  Non-Hispanic White | 43 | 46 | 89
  Black | 36 | 35 | 71
  Hispanic or Latino | 17 | 17 | 34
  Other | 5 | 4 | 9
Caregiver income (categorical) [Number; unit: participants]
  $<20,000 | 64 | 66 | 130
  $20,000-49,999 | 23 | 24 | 47
  $>=50,000 | 8 | 8 | 16
  Missing | 6 | 4 | 10
Patient income (categorical) [Number; unit: participants]
  $<20,000 | 37 | 46 | 83
  $20,000-49,999 | 49 | 44 | 93
  $>=50,000 | 7 | 6 | 13
  Missing | 8 | 6 | 14
Patient use of psychotropic medications (categorical) [Number; unit: participants]
  Yes | 5 | 8 | 13
  No | 96 | 93 | 189
  Missing | 0 | 1 | 1
Relationship of patient to his or her caregiver [Number; unit: participants]
  Spouse | 69 | 64 | 133
  Other family | 30 | 36 | 66
  Nonfamily | 2 | 2 | 4
Mini-blessed (continuous) [Mean (Standard Deviation); unit: units on a scale] — The mini-blessed measures cognitive impairment and responses to items are summed, resulting in a range of scores from 0 - 28, where higher scores indicate more cognitive impairment. Scores of 0-8 indicate no or minimal impairment, scores 9-19 indicate moderate impairment, and scores between 20-28 indicate severe impairment.
  units on a scale | 15.21 (7.36) | 14.70 (7.39) | 14.95 (7.36)
FAST stage (categorical) [Number; unit: participants] — The fast is a measure that ascertains which of the 7 stages of dementia one has: higher scores indicate more severe dementia. Stage 1 is normal adult with no functional decline, Stage 2 is normal older adult with some functional decline, Stage 3 is mild cognitive impairment, Stage 4 is mild dementia, Stage 5 is moderate dementia, Stage 6 is moderately severe dementia, and Stage 7 is severe dementia. Those with FAST scores between 2-6 were eligible for participation. We combined stages 2 and 3 (possible/mild cognitive impairment) and stages 5 and 6 (moderate/moderately severe dementia).
  participants
    Possible/mild cognitive impairment (stages 2-3) | 3 | 4 | 7
    Mild dementia (stage 4) | 23 | 24 | 47
    Moderate/moderately severe dementia (stages 5-6) | 74 | 73 | 147
    Missing | 1 | 1 | 2
Geriatric Depression Scale (continuous) [Mean (Standard Deviation); unit: units on a scale] — 30 item scale with response options of yes = 1 and no = 0 to each item. Total GDS scores range from 0 to 30, with greater scores indicating greater depression.
  units on a scale | 14.33 (6.22) | 13.97 (6.22) | 14.15 (6.21)
Enjoyment of Pleasant Events (continuous) [Mean (Standard Deviation); unit: units on a scale] — For each of 20 events, participants answered the frequency (0 = not at all, 1 = 1-6 times, 2 = 7+ times) they engaged in the event and whether they enjoyed the event (1 = yes, 0 = no). Scores for each of the 20 items were added together. The possible range of scores on the PES frequency of engagement in pleasant events is from 0 - 40, with higher scores indicating more frequent engagement in pleasant events.
  units on a scale | 23.09 (5.78) | 24.65 (7.39) | 23.87 (6.67)
Burden Severity (continuous) [Mean (Standard Deviation); unit: units on a scale] — 22 items are responded to on a 0-4 scale where 0 = never, 1 = rarely, 2 = sometimes, 3 = quite frequently, and 4 = nearly always. Scores are then summed so that the total range is from 0 - 88. Higher scores indicate greater caregiver burden.
  units on a scale | 28.94 (15.27) | 28.63 (15.18) | 28.78 (15.19)
Total Mutuality (continuous) [Mean (Standard Deviation); unit: units on a scale] — Fifteen items about the caregivers' relationship with the patient with dementia were responded to on a 0-4 scale, where 0 = not at all, 1 = a little, 2 = some, 3 = quite a bit, and 4 = a great deal. responses to all 15 items were averaged, so total scores range from 0-4, with higher values indicating greater mutuality.
  units on a scale | 2.93 (0.66) | 2.99 (0.66) | 2.96 (0.66)
Caregiver-reported Worst Pain (continuous) [Mean (Standard Deviation); unit: units on a scale] — One item with scores from 0 to 5, where 0 = no pain, 1 = little pain, 2 = moderate pain, 3 = quite bad pain, 4 = very bad pain, 5 = the pain is almost unbearable. Higher scores = greater pain severity.
  units on a scale | 3.28 (1.37) | 3.03 (1.29) | 3.15 (1.34)
Caregiver-reported Overall pain (continuous) [Mean (Standard Deviation); unit: units on a scale] — One item on a 0-5 scale, where 0 = no pain, 1 = little pain, 2= moderate pain, 3 = quite bad pain, 4 = very bad pain, 5 = the pain is almost unbearable. Higher scores = greater pain severity.
  units on a scale | 2.43 (1.13) | 2.06 (0.94) | 2.24 (1.05)
Patient-reported Worst pain (continuous) [Mean (Standard Deviation); unit: units on a scale] — One item on a 0-5 scale, where 0 = no pain, 1 = little pain, 2= moderate pain, 3 = quite bad pain, 4 = very bad pain, 5 = the pain is almost unbearable. Higher scores = greater pain severity.
  units on a scale | 3.01 (1.30) | 2.84 (1.51) | 2.93 (1.41)
Patient-reported Overall Pain [Mean (Standard Deviation); unit: units on a scale] — One item on a 0-5 scale, where 0 = no pain, 1 = little pain, 2= moderate pain, 3 = quite bad pain, 4 = very bad pain, 5 = the pain is almost unbearable. Higher scores = greater pain severity.
  units on a scale | 2.13 (1.11) | 1.96 (1.24) | 2.04 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Aggression as Determined by the Cohen-Mansfield Agitation Inventory (Aggression Subscale)
Description: The CMAI lists 13 behaviors (2 verbal and 11 nonverbal) and for each behavior the participant indicates how frequently the behavior occurs (1-5, higher values = greater frequency) and how disruptive the behavior is (1-5, higher values = greater disruptiveness). For any given behavior, if a participant scored a 2 or higher on BOTH frequency (i.e., it occurred "less than once a week" or more often) and disruptiveness (i.e., it was "a little" disruptive or more), he/she was considered aggressive.
  Overall aggression takes into account all 13 behaviors, whereas verbal aggression only pertains to two behaviors and non-verbal aggression pertains to 11 behaviors.
  One is considered verbally aggressive if he/she responds with a 2 or higher on both frequency and disruptiveness for either of the two verbal behaviors.
  One is considered non-verbally aggressive if he/she responds with a 2 or higher on both frequency and disruptiveness for any of the 11 non-verbal behaviors.
Time Frame: Three Months, Six Months, Twelve Months Post Intervention
Population: 203 community-dwelling Veterans with pain and dementia and their caregivers
Measure: Number; unit: participants
Groups:
- Arm 1: PAVeD Intervention: In the experimental arm, the caregiver will receive six to eight 45-minute visits to teach caregiver about pain and memory problems. The person with dementia will also be able to learn from these visits. These visits will take place over three months.
  PAVeD Intervention: In the PAVeD Intervention, the caregiver will receive six to eight 45-minute visits to teach caregiver about pain and memory problems. The person with dementia will also be able to learn from these visits. These visits will take place over three months. N = 101
- Arm 2: Enhanced Usual Care: In the comparison arm, the caregiver will receive information in the mail about memory problems and pain; and the caregiver will receive eight short telephone calls to check on how the person with dementia is doing.
  Enhanced Usual Care: In Enhanced Usual Care, the caregiver will receive information in the mail about memory problems and pain; and the caregiver will receive eight short telephone calls to check on how the person with dementia is doing.
  Primary Care providers will be notified through electronic medical records about any significant behavioral problems or pain.
  N = 102
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
participants
  3 month Overall Aggression | 8 | 14
  6 month Overal Aggression | 9 | 17
  12 month Overall Aggression | 17 | 14
  3 month Non-Verbal Aggression | 6 | 8
  6 month Non-Verbal Aggression | 5 | 6
  12 month Non-Verbal Aggression | 6 | 10
  3 month Verbal Aggression | 7 | 11
  6 month Verbal Aggression | 6 | 12
  12 month Verbal Aggression | 16 | 9
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Univariate time-to-event analyses, using discrete-time Cox regression models to evaluate differences between PAVeD and EU-PC in the primary outcome of incidence of aggression over time. We expected that patients with dementia among dyads randomized to PAVeD arm would be less likely to develop aggression compared to those randomized to the enhanced usual care arm; Test type: Non-Inferiority or Equivalence — Power calculations were based on the ability to detect a small-to-moderate difference (Cohen's h = .4) between treatment groups in rate of aggression onset over a 1-year period, assuming 80% power and T1 error rate of 5%. This differential rate in aggression onset is comparable to a 37% rate of aggression onset over a 1 year period for the control group versus 19% for the treatment group. Given this, our goal was to include 220 total participants (after 10% attrition: N = 198); p = 0.13, Regression, Cox — This is the p value from the discrete-time Cox regression time-to-event analyses; DF = 1; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.45 to 1.11] — The enhanced usual care arm is the comparison group
Statistical Analysis 2: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Comparison of incidence of non-verbal aggression between treatment groups; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.39, Regression, Cox — From discrete time-cox regression time-to-event analysis; df = 1; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.43 to 1.39] — The enhanced usual care arm is the reference group
Statistical Analysis 3: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Examination of group differences in incidence of verbal aggression. We expected those in paved to have lower incidence of verbal aggression relative to those in enhanced usual care; Test type: Non-Inferiority or Equivalence — Power calculations were based on the ability to detect a small-to-moderate difference (Cohen's h = .4) between treatment groups in rate of aggression onset (the primary outcome) over a 1-year period, assuming 80% power and type I error rate of 5%. This differential rate in aggression onset is comparable to a 37% rate of aggression onset over a 1 year period for the control group (anticipated based on estimated rates from prior work) versus 19% for the treatment group; p = 0.84, Regression, Cox — From discrete-time Cox regression time-to-event analyses; df = 1; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.51 to 1.37] — The usual care arm is the reference group

2. Secondary Outcome: Caregiver-Reported Worst Pain
Description: This is one item on the Philadelphia Pain Intensity Scale. One item with scores from 0 to 5, where 0 = no pain, 1 = little pain, 2 = moderate pain, 3 = quite bad pain, 4 = very bad pain, 5 = the pain is almost unbearable.
  Higher scores = greater pain severity
Time Frame: Baseline, 3 months, 6 months, and 12 months
Population: Growth curve models were conducted (n = 203) to examine whether there were treatment group differences in change over time in caregiver-reported worst pain.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 3.28 (1.37) | 3.03 (1.29)
  3 months | 2.83 (1.37) | 2.91 (1.40)
  6 months | 2.77 (1.39) | 2.85 (1.49)
  12 months | 2.70 (1.48) | 2.58 (1.39)
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Growth curve models were conducted to examine whether there were differences between treatment groups in change in caregiver reported worst pain over time; Test type: Superiority or Other; p = 0.46, Mixed Models Analysis — P value of the interaction between treatment group and time (time coded as 0, 3, 6, 12); F (3, 455) = 0.86; Results of F value of growth curve model = 0.86

3. Secondary Outcome: Patient-reported Worst Pain.
Description: This is one item on the Philadelphia Pain Intensity Scale. One item on a 0-5 scale, where 0 = no pain, 1 = little pain, 2= moderate pain, 3 = quite bad pain, 4 = very bad pain, 5 = the pain is almost unbearable.
  Higher scores = greater pain severity.
Time Frame: Baseline, 3, 6, and 12 months
Population: Growth curve models were conducted (n = 203) to examine whether there were treatment group differences in change over time in patient-reported worst pain.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 3.01 (1.30) | 2.84 (1.51)
  3 months | 2.49 (1.63) | 2.41 (1.62)
  6 months | 2.35 (1.54) | 2.72 (1.55)
  12 months | 2.54 (1.65) | 2.46 (1.81)
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.23, Mixed Models Analysis — P value of the interaction between treatment group and time (time coded as 0, 3, 6, 12); Results of F value of growth curve model = 1.43

4. Secondary Outcome: Caregiver Reported Overall Pain Over the Last Several Weeks
Description: as for outcome 3
Time Frame: Baseline, 3, 6, and 12 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 2.43 (1.13) | 2.06 (0.94)
  3 months | 1.99 (1.02) | 1.84 (0.99)
  6 months | 1.96 (1.13) | 1.96 (1.12)
  12 months | 2.00 (1.11) | 1.80 (1.08)
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Growth curve models were conducted to examine whether there were differences between treatment groups in change in caregiver reported overall pain over time; Test type: Superiority or Other; p = 0.23, Mixed Models Analysis — P value of the interaction between treatment group and time (time coded as 0, 3, 6, 12); F (3, 455) = 1.45; Results of F value of growth curve model = 1.45

5. Secondary Outcome: Patient-reported Overall Pain Over the Last Several Weeks
Description: as for outcome 3
Time Frame: Baseline, 3, 6, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 2.13 (1.11) | 1.96 (1.24)
  3 months | 1.71 (1.27) | 1.66 (1.37)
  6 months | 1.75 (1.25) | 1.92 (1.16)
  12 months | 1.77 (1.35) | 1.72 (1.40)
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Growth curve models were conducted to examine whether there were differences between treatment groups in change in patient-reported overall pain over time; Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — P value of the interaction between treatment group and time (time coded as 0, 3, 6, 12); F (3, 409) = 0.59; Results of F value of growth curve model = 0.86

6. Secondary Outcome: Depression
Description: Geriatric Depression Scale. 30 item scale with response options of yes = 1 and no = 0 to each item.
  Total GDS scores range from 0 to 30, with greater scores indicating greater depression.
Time Frame: Baseline, 3, 6, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 14.33 (6.22) | 13.97 (6.22)
  3 months | 13.17 (6.75) | 14.26 (6.96)
  6 months | 12.81 (6.82) | 14.01 (7.09)
  12 months | 13.12 (7.20) | 13.45 (7.53)
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Growth curve models were conducted to examine whether there were differences between treatment groups in change in depression over time; Test type: Superiority or Other; p = 0.42, Mixed Models Analysis — P value of the interaction between treatment group and time (time coded as 0, 3, 6, 12); F (3, 453) = 0.94; Results of F value of growth curve model = 0.94

7. Secondary Outcome: Pleasant Events - Short Form - Alzheimer's Disease
Description: The frequency of engagement in pleasant events, according to the Pleasant Events Schedule - Alzheimer's Disease.
  For each of 20 events, participants answered the frequency (0 = not at all, 1 = 1-6 times, 2 = 7+ times) they engaged in the event and whether they enjoyed the event (1 = yes, 0 = no).
  For each item, frequency x enjoyment were multiplied. Then scores for each of the 20 items were added together.
  The possible range of scores on the PES frequency of engagement in pleasant events is from 0 - 40, with higher scores indicating more frequent engagement in pleasant events.
Time Frame: Baseline, 0, 3, 6, 12 months
Population: Growth curve models were conducted (n = 203) to examine whether there were treatment group differences in change over time in frequency of pleasant events.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 23.09 (5.78) | 24.65 (7.39)
  3 months | 24.01 (6.31) | 24.81 (6.94)
  6 months | 24.41 (6.53) | 24.06 (7.50)
  12 months | 23.54 (6.51) | 2.74 (0.84)
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Growth curve models were conducted to examine whether there were differences between treatment groups in change in pleasant events over time; Test type: Superiority or Other; p = 0.35, Mixed Models Analysis — P value of the interaction between treatment group and time (time coded as 0, 3, 6, 12); F (3, 457) = 1.10; Results of F value of growth curve model = 1.10

8. Secondary Outcome: Caregiver Burden
Description: Caregiver-reported burden, according to the Burden Inventory. 22 items are responded to on a 0-4 scale where 0 = never, 1 = rarely, 2 = sometimes, 3 = quite frequently, and 4 = nearly always.
  Scores are then summed so that the total range is from 0 to 88. Higher scores indicate greater caregiver burden.
Time Frame: Baseline, 3, 6, 12 months
Population: Growth curve models were conducted (n = 203) to examine whether there were treatment group differences in change over time in caregiver burden.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 28.94 (15.27) | 28.63 (15.18)
  3 months | 26.88 (13.62) | 30.37 (16.88)
  6 months | 27.84 (16.48) | 32.00 (17.39)
  12 months | 27.46 (14.94) | 30.87 (16.18)
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Growth curve models were conducted to examine whether there were differences between treatment groups in change in caregiver burden over time; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis — P value of the interaction between treatment group and time (time coded as 0, 3, 6, 12); F (3, 456) = 2.00; Results of F value of growth curve model = 0.11

9. Secondary Outcome: Caregiver-perceived Mutuality
Description: Caregiver-Perceived Total Mutuality (with patient), based on the Mutuality Scale.
  Fifteen items about the caregivers' relationship with the patient with dementia were responded to on a 0-4 scale, where 0 = not at all, 1 = a little, 2 = some, 3 = quite a bit, and 4 = a great deal.
  responses to all 15 items were averaged, so total scores range from 0-4, with higher values indicating greater mutuality.
Time Frame: Baseline, 3, 6, 12 months
Population: Growth curve models were conducted (n = 203) to examine whether there were treatment group differences in change over time in caregiver-reported mutuality.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 2.93 (0.66) | 2.99 (0.66)
  3 months | 3.01 (0.69) | 2.82 (0.80)
  6 months | 3.02 (0.64) | 2.78 (0.79)
  12 months | 2.82 (0.72) | 2.74 (0.84)
Statistical Analysis 1: Comparison: Arm 1: PAVeD Intervention vs Arm 2: Enhanced Usual Care; Growth curve models were conducted to examine whether there were differences between treatment groups in change in caregiver reported mutuality over time; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — P value of the interaction between treatment group and time (time coded as 0, 3, 6, 12); F (3, 456) = 3.84; Results of F value of growth curve model = 3.84

ADVERSE EVENTS:
Time Frame: Throughout the study; during sessions and assessments (3, 6, and 12 months)
Arm/Group | Arm 1: PAVeD Intervention | Arm 2: Enhanced Usual Care
Serious Adverse Events (participants affected / at risk) | 6/101 | 13/102
Other Adverse Events (participants affected / at risk) | 0/101 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: PAVeD Intervention (N=101) | Arm 2: Enhanced Usual Care (N=102)
Deceased - Unrelated to Study (General disorders) | 6 (6) | 13 (13) — We cannot specify why these people passed away.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes